CLINICAL TRIAL: NCT01744639
Title: Analysis of Body Composition by Bioelectrical Impedance in Patients With Hepatocellular Carcinoma (HCC) Undergoing Treatment Radioablation
Brief Title: Analysis of Body Composition in Patients With Hepatocellular Carcinoma in Radioablation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to find patients
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, ALDO TORRE DELGADILLO, Investigador Principal, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GAS 720-12/13-1
Record Dates: First submitted 2012-12-05; First posted 2012-12-07 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Liver Carcinoma
Keywords: Hepatocellular carcinoma; Radioablation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Anthropometry; Electric Impedance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HCC under treatment with radioablation (Experimental): Assessment of nutritional status by anthropometry, bioelectrical impedance, blood sampling and application of psychometric hepatic encephalopathy score and critical flicker frequency, to assess the presence of hepatic encephalopathy.
  Interventions: Behavioral: HCC under treatment with radioablation

INTERVENTIONS:
Behavioral: HCC under treatment with radioablation — The evaluation will take place over a period of 30 days.
  Other Names: Anthropometry; Bioelectrical impedance

SUMMARY:
Number of shows: 20 patients Track: A month with three visiting Intervention: Nutritional assessment including anthropometry, bioelectrical impedance, biochemical tests, Psychometric Hepatic Encephalopathy Score and Critical Flicker Frequency.

DETAILED DESCRIPTION:
There will be a prospective, longitudinal, comparative. It included 20 patients diagnosed with hepatocellular carcinoma. As there are a finite number of active patients at the institute, and no studies with sample size well established, has seen a sample size of 20 patients.

The duration of individual monitoring shall be one month to three visits (baseline, week 2 and week 4 after receiving the first radiofrequency ablation). Each visit will be a nutritional assessment including anthropometry, bioelectrical impedance, biochemical tests, Psychometric Hepatic Encephalopathy Score (PHES) and Critical Flicker Frequency (CFF).

Anthropometric measures to be taken are weight, height and arm circumference average.

Bioelectrical impedance will be using a single frequency impedance meter (425 to -50 KHz, Range 0 to 10,000) Bioelectrical Body Composition Analyzer Quantium II RJL Systems. The team measured the subjects' impedance, resistance, reactance and phase angle by Lean Body program provided by the manufacturer.

Hepatic encephalopathy be evaluated by testing PHES and was measured CFF, also also be measured ammonium, tumor necrosis factor, IL-1, IL-6, IL-10, renin angiotensin aldosterone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of hepatocellular carcinoma, treatment-naive and who are referred to the radiology department for radioablation as first therapy.
* Outpatients.
* Willingness to participate in the project.

Exclusion Criteria:

* Patients with hepato-renal diseases.
* Patients diagnosed with hepatocellular carcinoma undergoing chemoembolization treatment, or who have received more than one session radioablation.
* Patients with depression or psychiatric illnesses
* Patients who do not agree to participate in the project.

Exclusion Criteria:

* incomplete Applied Tests
* disagreement of the person to perform any of the tests
* monitoring Breach
* Hospitalization or death after the first session radioablation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Nutritional Status | Participants will be evaluated for a month
  Measured with the following parameters:body weight and height (to calculate BMI), triceps skinfold and mid-arm circumference (to calculated mid-arm muscle circumference, fat mass, fat free mass total, intracellular and extracellular body water obtained by bioelectrical impedance analysis and individual vectors obtained by bioelectrical impedance vector analysis.

SECONDARY OUTCOMES:
Minimal hepatic encephalopathy | Participants will be assessed for one month
  Assessed by psychometric Hepatic Encephalopathy (PHES) and Critical Flicker Frequency (CFF)

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Torre Delgadillo, M.D. M.Sc, Principal Investigator — INCMNSZ
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, D.f., Mexico